CLINICAL TRIAL: NCT01673906
Title: Accuracy and Clinical Impact of 68-Ga-labeled Octreotide Analogues PET in Diagnosis and Staging of Duodenal-pancreatic Neuroendocrine Tumours; Proposal of a Multicenter, Prospective Clinical Trial
Brief Title: 68-Ga-labeled Octreotide Analogues PET in Duodenal-pancreatic Neuroendocrine Tumours
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2012-000994-22; 2012-000994-22 (EudraCT Number)
Record Dates: First submitted 2012-08-09; First posted 2012-08-28 (Estimated); Last update posted 2025-06-24 (Actual); Status verified 2018-03

CONDITIONS: Neuroendocrine Tumours
Keywords: positron-emission tomography; neuroendocrine tumors; endosonography; tomography, X-ray computed; biopsy, fine needle; sensitivity and sensibility
MeSH Terms: conditions — Neuroendocrine Tumors; Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic work up (Experimental): The patients enrolled in the study (see below), with a consistent clinical suspicion of a primary duodenal-pancreatic NET.
  Interventions: Drug: Diagnostic work up

INTERVENTIONS:
Drug: Diagnostic work up — Patients will undergo MDCT, PET and EUS. Every attempt will be made to achieve a pre-operative cytologic diagnosis of any primary lesion by EUS-FNA. All diagnostic tests (MDCT, PET, EUS) should be performed during a two month time span, in this fixed order. The nuclear medicine doctor will be blinded of findings of MDCT. The gastroenterologist will be blinded about the findings of MDCT and PET until he has completed the diagnostic EUS. For ethical reasons, the findings of MDCT and PET will be disclosed to her/him, while the patient is still sedated in the operating room, just before the FNA. The minimal technical requirement for the techniques, the requested levels of clinical competence of the operators and the procedure for critical revision of radiological and cytological and histological specimens are detailed in the protocol. For PET any 68Ga -labeled-octreotide analogue will be allowed. Before EUS, an extended-esophagogastroduodenoscopy (until the Treitz) until will be performed.

SUMMARY:
The diagnostic work-up of patients suspected of having neuroendocrine tumours (NETs) has traditionally been a challenging issue. The last two decades have been marked by the application to use in the diagnosis of NETs of 3 newly available diagnostic techniques: endoscopic ultrasonography (EUS), multidetector CT (MDCT), and more recently, positron emission tomography using 68Ga-labelled octreotide analogues (PET). In a prospective study conducted at a single referral centre that compared PET with conventional somatostatin receptor scintigraphy and MDCT in diagnosis, staging and follow-up of patients affected by NET, PET detected more primary and secondary lesions than other methods. Recent studies investigated the clinical impact of PET in the management of patients affected by NET, previously studied by MDCT. The investigators recently reported the results of the investigation of 19 patients suspected of having primary pancreatic NET and studied by PET, MDCT and EUS. The investigators preliminary data suggest that PET may be slightly more sensitive than MDCT in detecting small (<2cm) pancreatic lesions; accuracy of PET and EUS is probably similar. No prospective study has yet been devoted to evaluate the accuracy of PET in the diagnosis and staging of primary duodenal-pancreatic NETs. Furthermore, the clinical impact of the adjunct of PET to the traditional protocols of diagnosis and staging of these tumours waits to be thoroughly evaluated. Thus the appropriate place of PET in the diagnostic algorithm of patients suspected of having duodenal-pancreatic NET remains undefined.

The main aim of this project is to prospectively compare the accuracy of PET and MDCT in the diagnosis and staging of patients suspected of having duodenal-pancreatic NETs. The investigators hypothesised that PET is superior to MDCT in the diagnosis of these neoplasm (the dimension of the study sample is estimated in order to detect a 10% difference). The impact of PET on management plan of affected patients will also be evaluated. As a secondary endpoint of the study, the investigators will compare EUS, PET and MDCT in the diagnosis of primary duodenal-pancreatic NET. The study is designed as a multicentre, prospective, non-randomised clinical trial. All patients will undergo MDCT, PET and EUS in this fixed order.

ELIGIBILITY:
Inclusion Criteria:

1. Patients affected by proved MEN-I, in whom a neoplasm in the duodenal-pancreatic area is suspected.
2. Patients with clinical diagnosis of carcinoid syndrome.
3. Patients with clinical diagnosis of Zollinger-Ellison syndrome.
4. Patients with insulinoma, as proved by fasting test.
5. Patient with clinical pictures and laboratory findings suggesting other functional or non-functional NET.
6. Patients who had previously undergone surgery, including total and subtotal pancreatectomy, or a duodenotomy, intended as curative for a histologically confirmed NET.
7. Patients who were diagnosed with NET metastasis with unknown primary location of the disease.
8. Patients undergoing diagnostic work-up for a periduodenal or pancreatic lesion incidentally found during abdominal ultrasound (not performed for suspicion of a NET) and with ultrasonographic characteristics (rounded, hypoechoic or egg-eye, well demarcated) suspicious for NET.
9. Patients undergoing diagnostic work-up for a periduodenal or pancreatic lesion incidentally found during TC (not performed for suspicion of a NET) and with radiological characteristics (well demarcated, hypervascular) suspicious for NET.

Exclusion criteria:

1. Patient unwilling, or unable to consent.
2. Pregnancy, or lactation.
3. Age <18 years
4. Known diagnosis of duodenal-pancreatic NET.
5. Patients with concomitant life-threatening disease.
6. Patients who had already undergone PET or EUS, in the last six months. In particular patients should be excluded from the study, when a lesion in the duodenal-pancreatic area, with characteristic suspicious for a NET, is incidentally diagnosed by PET, or EUS, or when a previously unsuspected diagnosis of NET is suggested by EUS-FNA of a pancreatic lesion.
7. Patients who had previously undergone total gastrectomy or pancreatectomy will be included in the study, but they will not undergo EUS.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2012-08; Primary Completion 2015-08 (Actual); Study Completion 2016-07-05 (Actual)

PRIMARY OUTCOMES:
Accuracy of the diagnostic test. | one year
  Accuracy was computed as: (number of true positives + true negatives)/(number + true positives + true negatives + false positives + false negatives). Accuracy of MDCT and PET in the diagnosis of primary duodenal-pancreatic NET will be calculated on a patient basis and they will be compared using McNemar test. Reference standard will be considered the diagnoses of primary NET, when supported by unambiguous cytology, histology or by at least one year of follow up.In cases of disagreement between cytological and histological findings, histology will be the gold standard.
Accuracy of the diagnostic test (after exclusion of patients enrolled due to a incidentally diagnosed lesion) | one year
  Accuracy was calculated as above, but based on subjects matching criteria 1-7 of the list of clinical situations suggestive for NET (see below, inclusion criteria). Patients with a lesion suspicion of NET incidentally diagnosed during abdominal ultrasound or MDCT not performed for clinical suspicion of NET were excluded.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety. | one year
  Number of patients with adverse events of each procedure: PET, MDCT, endoscopic ultrasonography-fine needle aspiration (EUS-FNA)
Sensitivity of the diagnostic tests. | one year
  Sensitivity (Number of true positive results/number of true positive + false negative results) of the diagnostic tests in the diagnosis of primary duodenal-pancreatic NET. Sensitivity of each diagnostic test (MDCT, PET, EUS) will be calculated separately on patient (number of true affected patients/number of true affected + number of false non affected patients) and on lesion basis (number of true positive lesions/number of true positive + false positive lesions)with its 95% confidence interval based on normal approximation.Reference standard will be considered the diagnoses of primary NET, when supported by unambiguous cytology, histology or by at least one year of follow up.In cases of disagreement between cytological and histological findings, histology will be the gold standard.
Specificity of the diagnostic tests. | one year
  Specificity (Number of true negative results/number of true negative + false positive results) of the diagnostic tests in the diagnosis of primary duodenal-pancreatic NET. Specificity of each diagnostic test (MDCT, PET, EUS) will be calculated separately on patient (number of true non affected patients/number of true non affected + number of false affected patients) and on lesion basis (number of true negative lesions/number of true negative positive + false positive lesions)with its 95% confidence interval based on normal approximation.Reference standard will be considered the diagnoses of primary NET, when supported by unambiguous cytology, histology or by at least one year of follow up.In cases of disagreement between cytological and histological findings, histology will be the gold standard.
Clinical impact of PET. | one year
  Changes in management plan in consequence of PET results. Prior to receiving the results of the PET scans, the referring clinician will be required to explicit a management plan for the patient. Following the release of the PET results, a second management plan will be recorded, including any changes resulting from the PET findings. The number of patients with changes in their management plan will be recorded.
Diameter of lesions. | one year
  Median diameter (cm) and ranges of lesions diagnosed by each technique will be calculated.

OTHER OUTCOMES:
Accuracy of EUS-FNA | one year
  Accuracy was computed as: (number of true positives + true negatives)/(number + true positives + true negatives + false positives + false negatives). Reference standard will be considered the diagnoses of primary NET, when supported by histology or by at least one year of follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Camellini, MD, Study Director — Gastroenterology and Digestive Endoscopy Unit, Santa Maria Hospital, Reggio Emilia, Italy.; Gabriele Carlinfante, MD, Study Director — Unit of Pathology, Santa Maria Nuova Hospital, Reggio Emilia, Italy; Andrea Frasoldati, MD, Study Director — Department of Endocrinology, Thyroid Disease Center-Arcispedale Santa Maria Nuova of Reggio Emilia, Reggio Emilia, Italy.; Armando Froio, Biologist, Study Director — Nuclear Medicine Unit, Santa Maria Nuova Hospital; Tiziana Cassetti, Biologist, Study Director — Gastroenterology and Digestive Endoscopy Unit, Santa Maria Hospital, Reggio Emilia, Italy.
Locations (21):
- Irene Virgolini, Innsbruck, Innsbruck, Austria
- Italy (20):
  - Nadia Cremonini, Bologna, Bologna
  - Fernando Cirillo, Cremona, Cremona
  - Diego Ferone, Genova, Genova
  - Giovanna Pepe, Milan, Milano
  - Rita Conigliaro, Modena, Modena
  - Luppi Gabriele, Modena, Modena
  - Pellegrino Crafa, Parma, Parma
  - Piero Ferolla, Perugia, Perugia
  - Antonio Chella, Pisa, Pisa
  - Laura Scaltriti, Guastalla, Reggio Emilia
  - ASMN IRCCS Reggio Emilia, Reggio Emilia, RE
  - Enrico Papini, Albano Laziale, Roma
  - Roberto Baldelli, Roma, Roma
  - Vittoria Rufini, Roma, Roma
  - Claudio De Angelis, Torino, Torino
  - Marco Gallo, Torino, Torino
  - Paolo Limone, Torino, Torino
  - Franco Grimaldi, Udine, Udine
  - Massimo Falconi, Verona, Verona
  - Roberto Castello, Verona, Verona

REFERENCES:
- [Background] Gabriel M, Decristoforo C, Kendler D, Dobrozemsky G, Heute D, Uprimny C, Kovacs P, Von Guggenberg E, Bale R, Virgolini IJ. 68Ga-DOTA-Tyr3-octreotide PET in neuroendocrine tumors: comparison with somatostatin receptor scintigraphy and CT. J Nucl Med. 2007 Apr;48(4):508-18. doi: 10.2967/jnumed.106.035667. PMID 17401086
- [Background] Ambrosini V, Campana D, Bodei L, Nanni C, Castellucci P, Allegri V, Montini GC, Tomassetti P, Paganelli G, Fanti S. 68Ga-DOTANOC PET/CT clinical impact in patients with neuroendocrine tumors. J Nucl Med. 2010 May;51(5):669-73. doi: 10.2967/jnumed.109.071712. Epub 2010 Apr 15. PMID 20395323
- [Background] Versari A, Camellini L, Carlinfante G, Frasoldati A, Nicoli F, Grassi E, Gallo C, Giunta FP, Fraternali A, Salvo D, Asti M, Azzolini F, Iori V, Sassatelli R. Ga-68 DOTATOC PET, endoscopic ultrasonography, and multidetector CT in the diagnosis of duodenopancreatic neuroendocrine tumors: a single-centre retrospective study. Clin Nucl Med. 2010 May;35(5):321-8. doi: 10.1097/RLU.0b013e3181d6677c. PMID 20395703